CLINICAL TRIAL: NCT05771415
Title: Near-infrared Spectroscopy: Differences in Placental Oxygenation in Relation to Ultrasound Maturation Grade in physiologIcal Term Pregnancies
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Andrea Etrusco, Principal investigator, University of Palermo
Other Study IDs: PLA-OX-1
Record Dates: First submitted 2023-02-08; First posted 2023-03-16 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Placenta Diseases
Keywords: Near-Infrared Spectroscopy; Placenta oxigenations; Placenta maturity
MeSH Terms: conditions — Placenta Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Grannum placental maturity grade 0 and 1 (low maturity level: Women with low placental maturity grade (group 1, Grannum 0-1)
- Grannum placental maturity grade 2 and 3 (high maturity level): Women with high placental maturity grade (group 2, Grannum 2-3)

SUMMARY:
The aim was to compare placental oxygenation in low risk, uncompli-cated, term pregnancies measured by near-infrared spectroscopy (NIRS) in relation to the placental maturity grade determined by ultrasound assessment according to Grannum scale.

The study included 34 singleton subjects divided into two groups accord-ing to placental maturation: low grade (Grannum 0-1; n=10) and high grade (Gran-num 2-3; n=24). In each study subjects, measurement was performed at two sites: (a) test site above the central part of the placenta, and (b) control site out of placenta on lower abdomen, in medial line, 3 cm from the symphysis. Student's t-test was used to compare tissue oxygenation index (TOI) values among the study groups. The normality of distribution was demonstrated by the Kolmogorov-Smirnov test.

ELIGIBILITY:
Inclusion Criteria:

singleton pregnancies low-risk pregnancies uncomplicated pregnancies term pregnancies (37th to 41+6 weeks of gestation) anterior placental localization abdominal wall of less than 3cm thickness.

Exclusion Criteria:

complicated pregnancies pre-term pregnancies Abdominal wall tick > 3cm

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: pregnant women with singleton low-risk, uncomplicated, term pregnancies anterior placental localization and abdominal wall of less than 3cm thickness. US and Doppler studies, as well as CTG and laboratory findings were normal in all study women.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Placental oxygenation levels | During the procedure
  to compare placental oxygenation in low risk, uncomplicated, term pregnancies measured by near-infrared spectroscopy (NIRS) in relation to the placental maturity grade determined by ultrasound assessment according to Grannum scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mislav Mikuš, M.D., Principal Investigator — Clinical Hospital Centre Zagreb; Antonio Simone Laganà, M.D. Ph.D., Study Chair — University of Palermo; Andrea Etrusco, M.D, Study Chair — University of Palermo
Locations (1):
- Hormona Polyclinic, Split, Croatia